CLINICAL TRIAL: NCT07123844
Title: The Effects of Cholesterol-Restricted Diets Enriched With Pumpkin Seeds and Pumpkin Seed Oil on Cardiovascular Risk Factors in Individuals With Hyperlipidaemia
Brief Title: Pumpkin Seeds or Oil Lower Serum Triglyceride Levels in Individuals With Hyperlipidaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Collaborators: Okan University (Other)
Responsible Party: Principal Investigator, Kevser Karli, Principal Investigator, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022--KAEK-37
Record Dates: First submitted 2025-07-30; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hyperlipidemia; Overweight
Keywords: overweight; pumpkin seed; pumpkin seed oil; nutritional treatment; functional food; hyperlipidemia; serum lipids
MeSH Terms: conditions — Hyperlipidemias; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pumpkin seed (Experimental): 30 g/day pumpkin seed and low cholesterol diet (28 days)
  Interventions: Dietary Supplement: low cholesterol diet
- pumpkin seed oil (Experimental): 15 g/day pumpkin seed oil and low cholesterol diet (28 days)
  Interventions: Dietary Supplement: low cholesterol diet
- control (Experimental): low cholesterol diet (28 days)
  Interventions: Dietary Supplement: low cholesterol diet

INTERVENTIONS:
Dietary Supplement: low cholesterol diet — low cholesterol diet

SUMMARY:
Aim of the Study:

This randomized controlled experimental study aimed to evaluate the effects of cholesterol-restricted diets enriched with pumpkin seeds and pumpkin seed oil on cardiovascular risk factors-specifically serum lipid profile (total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides), blood pressure, and anthropometric measurements (body weight, body mass index, body fat percentage, and fat mass)-in individuals with hyperlipidemia.

Research Questions:

Does the nutritional intervention lead to a reduction in serum total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), and triglyceride (TG) levels, as well as an increase in high-density lipoprotein cholesterol (HDL-C) levels across all study groups?

Do the groups receiving diets enriched with pumpkin seeds or pumpkin seed oil show greater improvements in lipid profile (TC, LDL-C, TG) and a more pronounced increase in HDL-C compared to the control group?

Does the nutritional intervention result in reductions in body weight, BMI, body fat percentage, and fat mass in all study groups?

DETAILED DESCRIPTION:
The aim of this randomized controlled trial was to investigate the effects of cholesterol-restricted diets enriched with pumpkin seeds or pumpkin seed oil on cardiovascular risk factors in individuals with hyperlipidemia. Specifically, the study aimed to determine the effects of these dietary interventions on serum lipid parameters (total cholesterol, LDL-cholesterol, HDL-cholesterol, and triglycerides), blood pressure (systolic and diastolic), and anthropometric measurements (body weight, body mass index, body fat percentage, and fat mass) over a 28-day period.

The study hypothesizes that incorporating pumpkin seeds or pumpkin seed oil into a cholesterol-restricted diet will improve serum lipid parameters and blood pressure, and reduce anthropometric measurements.

Research Questions:

Primary Questions:

Does consumption of a cholesterol-restricted diet in individuals with hyperlipidemia result in statistically significant improvements in the serum lipid profile (i.e., decreases in TC, LDL-C, and TG, and increases in HDL-C)?

Do diets enriched with pumpkin seeds or pumpkin seed oil lead to greater improvements in these lipid parameters compared to a control group that only follows a cholesterol-restricted diet?

Secondary Questions:

Does the intervention (regardless of group) lead to reductions in anthropometric indices such as body weight, BMI, body fat percentage, and fat mass?

Are reductions in anthropometric measurements and improvements in blood pressure more pronounced in groups consuming diets enriched with pumpkin seeds or pumpkin seed oil compared to the control group?

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria:

* Aged between 19 and 64 years
* Body mass index (BMI) between 25.0 and 30.0 kg/m²
* Triglyceride (TG) level > 200 mg/dL
* Low-density lipoprotein cholesterol (LDL-C) between 130 and 190 mg/dL
* Fasting blood glucose < 110 mg/dL
* Blood pressure below 140/90 mmHg

Exclusion Criteria

* Individuals will be excluded if they meet any of the following criteria:
* Diagnosis of any systemic disease, including:
* Diabetes mellitus
* Hypertension
* Cancer
* Metabolic syndrome
* Chronic kidney disease
* Use of any medication that affects blood lipid, glucose, and pressure levels
* Presence of food allergies (e.g., to pumpkin seeds or oil)
* Current or recent nutritional treatment or dietary therapy
* Pregnancy or breastfeeding
* Diagnosed psychiatric disorders
* Known congenital metabolic disorders

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Change in Serum Total Cholesterol (mg/dL) from Baseline to Day 28 | Baseline and Day 28
  Measured from 12-hour fasting venous blood samples using enzymatic colorimetric methods on an automated analyzer. Reference ranges per Turkish Society of Endocrinology and Metabolism (TEMD) Dyslipidemia Guidelines, 2021: desirable <200 mg/dL, borderline high 200-239 mg/dL, high ≥240 mg/dL.
Change in Serum LDL-Cholesterol (mg/dL) from Baseline to Day 28 | Baseline and Day 28
  Calculated using the Friedewald formula from fasting lipid profile. Reference ranges per TEMD, 2021: optimal <100 mg/dL (or <70 mg/dL for very high cardiovascular risk), borderline high 130-159 mg/dL, high 160-189 mg/dL, very high ≥190 mg/dL.
Change in Serum HDL-Cholesterol (mg/dL) from Baseline to Day 28 | Baseline and Day 28
  Measured from fasting venous blood using enzymatic methods. Reference ranges per TEMD, 2021: low HDL <40 mg/dL in men and <50 mg/dL in women; protective ≥60 mg/dL.
Change in Serum Triglycerides (mg/dL) from Baseline to Day 28 | Baseline and Day 28
  Measured from fasting venous blood using enzymatic methods. Reference ranges per TEMD, 2021: normal <150 mg/dL, borderline high 150-199 mg/dL, high 200-499 mg/dL, very high ≥500 mg/dL.

SECONDARY OUTCOMES:
Change in Body Weight (kg) from Baseline to Day 28 | Baseline and Day 28
  Measured without shoes and in light clothing using a Tanita TBF-300 bioelectrical impedance analyzer (BIA).
Height (m) at Baseline | Baseline
  Measured using a Densi GL 150 stadiometer.
Change in Body Mass Index (kg/m²) from Baseline to Day 28 | Baseline and Day 28
  Calculated as body weight (kg) divided by height squared (m²). Classification per World Health Organization (WHO): normal 18.5-24.9, overweight 25.0-29.9, obese ≥30.0.
Change in Body Fat Percentage (%) from Baseline to Day 28 | Baseline and Day 28
  Measured using a Tanita TBF-300 BIA.
Change in Fat Mass (kg) from Baseline to Day 28 | Baseline and Day 28
  Measured using a Tanita TBF-300 BIA.
Change in Systolic Blood Pressure (mmHg) from Baseline to Day 28 | Baseline and Day 28
  Measured in seated position after 5 minutes of rest using an automated sphygmomanometer. Two readings taken 1-2 minutes apart; average recorded. Reference ranges per ESC/ESH Guidelines, 2018: normal <120 mmHg; elevated 120-139 mmHg.
Change in Diastolic Blood Pressure (mmHg) from Baseline to Day 28 | Baseline and Day 28
  Same procedure as systolic BP measurement. Reference ranges per ESC/ESH Guidelines, 2018: normal <80 mmHg; elevated 80-89 mmHg.
Change in Dietary Energy and Nutrient Intake (kcal/day, g/day, mg/day) from Baseline to Day 28 | Baseline and Day 28
  Assessed by 3-day food records (two weekdays and one weekend day). Data analyzed using the Nutrition Information System (BeBİS, version 7.2). Results compared with recommended daily intakes in the Turkish Nutrition Guide (TÜBER, 2022).
Change in Food Group Consumption Frequency (times/week) from Baseline to Day 28 | Baseline and Day 28
  Evaluated using a structured dietary habits questionnaire. Frequency data categorized by major food groups and analyzed for change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Öngün Yılmaz, pHD, Study Director — hyilmaz@bandirma.edu.tr
Locations (1):
- Kastamonu Training and Research Hospital, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and informed consent form will be shared with other researchers upon request. However, no individual participant data (IPD) such as de-identified participant-level health data will be shared. The shared documents will not include any personal or outcome data of participants.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 6 months after the publication of the main study results.
Access Criteria: Interested researchers may request access by contacting the investigator via email at kevserkarli@gmail.com or kevserkarli@kastamonu.edu.tr. Data will be shared via secure email format.